CLINICAL TRIAL: NCT07120334
Title: mHealth Dietary Intervention for Stroke Survivors With Prediabetes or T2D
Brief Title: Mobile Health Dietary Intervention for Stroke Survivors With Prediabetes or Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Queen's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RA-2025-302
Record Dates: First submitted 2025-07-28; First posted 2025-08-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stroke Recurrence; Type 2 Diabetes; Prediabetes
Keywords: PortionSize Ed; Stroke; Diabetes; Prediabetes; Type 2 Diabetes; T2D; Mediterranean Diet; mHealth; Hawaii
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Stroke; Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PortionSize Ed + MedDiet Support (Experimental): Full PortionSize Ed app access with personalized dietary feedback, educational videos, 3 virtual sessions with a registered dietitian (RDN), standard of care (for post-stroke with pre-diabetes or T2D) over 12 weeks.
  Interventions: Behavioral: PortionSize Ed + MedDiet Support
- Standard of Care (Active Comparator): Uses a basic version of the app without feedback or RDN support and receives usual care for stroke recovery for 12 weeks.
  Interventions: Behavioral: Standard of care for Stroke and Prediabetes or T2D

INTERVENTIONS:
Behavioral: PortionSize Ed + MedDiet Support — Full PortionSize Ed app access with personalized dietary feedback, educational videos, 3 virtual sessions with a registered dietitian (RDN), standard of care (for post-stroke with pre-diabetes or T2D) over 12 weeks.
  Arms: PortionSize Ed + MedDiet Support
Behavioral: Standard of care for Stroke and Prediabetes or T2D — Uses a basic version of the PortionSize Ed app without feedback or RDN support and receives usual care for stroke recovery and prediabetes or T2D for 12 weeks.
  Arms: Standard of Care

SUMMARY:
Objectives: This study aims to test whether a mobile app called PortionSize Ed can help adults who have had a recent stroke and also have prediabetes or type 2 diabetes improve their diet. Specifically, we want to see if the app can help people follow a Mediterranean-style diet, which may lower the risk of future strokes and improve overall health.

The main goals are to:

* Test if the app is easy to use and acceptable to participants.
* See whether the app helps people follow a healthier diet.
* Look at changes in health indicators like blood sugar, cholesterol, blood pressure, and body fat.

Design and Outcome:

This is a randomized controlled pilot study that will involve 40 participants. All participants will be recruited from Queen's Medical Center after a recent stroke and will be randomly assigned to one of two groups:

Intervention Group: Uses the full PortionSize Ed app, gets weekly reminders and educational videos, and has 3 sessions with a registered dietitian (RDN) over 12 weeks.

Control Group: Uses a basic version of the app without feedback or RDN support, and receives usual care for stroke recovery.

All participants will continue to receive standard care from Queen's, including the My Stroke Recovery Guide. The study lasts 12 weeks, with visits at the beginning and end to collect health data and feedback on the app.

Schedule and Type of Evaluations/Interventions:

Participants will complete the following:

Baseline and Week 12 Visits: In-person assessments for blood sugar (HbA1c), cholesterol, blood pressure, height, weight, and body composition (using DXA, BIA, and 3D imaging), as well as surveys about their diet and activity levels.

Intervention Group Only:

* Three virtual counseling sessions with a registered dietitian (Week 1, 6, 12)
* Weekly nutrition goal tracking and texting with the dietitian
* Watching short educational videos through the app
* Receiving app-based feedback on how well their diet follows Mediterranean Diet recommendations

Duration of Study: The study will last 12 weeks for each participant, with an optional long-term follow-up using medical records.

Sample Size and Population: The study will include 40 adults, ages 30 to 65, who:

* Recently experienced a stroke
* Have a history of prediabetes or type 2 diabetes
* Are medically stable and able to use a smartphone (or willing to use a study-provided iPhone)
* People will be excluded if they have severe swallowing issues, cognitive problems, or dietary needs that would make it hard to follow a Mediterranean-style diet.

DETAILED DESCRIPTION:
Study Visits:

Baseline Visit (Week 0) at UHCC - All Participants:

* Consent form signed and randomization to a study group
* Fingerstick blood test to measure HbA1c and lipid levels
* Height, weight, blood pressure, and body composition measurements using DXA, BIA, and 3D Optical Scan
* Questionnaires: Demographics, physical activity (IPAQ-SF), Mediterranean Diet adherence (MEDAS), and current medications
* PortionSize Ed app training and 3-day food logging using the app
* Pregnancy test (urine) for participants of childbearing potential
* Counseling with the registered dietitian (~30-60 minutes) (Intervention only)
* Receive study stipend ($50)

Week 6 Visit, Virtual Visit:

* Follow-up questionnaires and review of app engagement (Intervention only)
* Counseling with the registered dietitian (~30-60 minutes) (Intervention only)
* Review of medications and dietary services received
* Self-reported adherence and barriers to diet change (Intervention only)
* Receive study stipend ($60)

Week 12 Visit at UHCC - All Participants:

* Repeat body composition measurements (DXA, BIA, 3DO)
* Repeat fingerstick blood tests (HbA1c and lipids)
* Final questionnaires and MEDAS
* Final 3-day food record
* Satisfaction and usability surveys
* Counseling with the registered dietitian (~30-60 minutes) (Intervention only)
* Return study iPhone (if applicable)
* Receive study stipend ($90)

Between visits for intervention group only:

* Log one day food intake per week (~10-15 minutes)
* Text weekly dietary goal (~5 minutes)
* Watch a short nutrition video each week (~3 minutes)
* Weekly reminders to complete a 1-day food log/week between study visits

Between visits for Active Comparator Group:

• Basic version of the app (no real-time feedback or counseling) and continue usual care, including the My Stroke Recovery Guide.

Length of Time in this Study:

Participation in this study will last approximately 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 to 65 years
* Recent stroke (ischemic, hemorrhagic or Transient Ischemic Attack), within 1-14 days prior to enrollment
* Confirmed diagnosis of prediabetes or type 2 diabetes, based on HbA1c results
* Medically stable and cleared for oral diet and physical activity by the attending physician
* Cleared for thin liquids and regular textures by physician
* Capable of providing informed consent
* Able to speak and read English
* Owns a smartphone OR is willing to use a study-provided iPhone
* Has sufficient cognitive and physical function to use a mobile app
* Willing to participate in all study procedures and available for the 12-week duration

Exclusion Criteria:

* Severe dysphagia that prevents oral intake
* Type 1 diabetes
* Cognitive impairment (e.g., dementia, post-stroke confusion) that precludes consent or compliance, as judged by the clinical care team
* Current participation in another interventional clinical trial
* Pregnant or breastfeeding, or planning to become pregnant during the study period
* Unwilling or unable to provide written informed consent
* Serious comorbid conditions that, in the opinion of the

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant Acceptability of PortionSize Ed App | 11 months
  Mean acceptability score measured by the Computer System Usability Questionnaire (CSUQ), a validated 19-item Likert scale instrument assessing system usefulness, information quality, and interface quality. Each item is scored on a 7-point scale ranging from 1 (Strongly Agree) to 7 (Strongly Disagree).
  Unit of Measure: Mean CSUQ score (1-7) Direction of Scoring: Lower scores indicate higher acceptability and better usability.
Participant Retention Rate | 11 months
  Percentage of participants who complete all scheduled study assessments (Weeks 1, 6, 12). Higher percentages indicate better retention and feasibility of the intervention.
Participant Satisfaction with Study Procedures and App Features | 11 months
  Description:
  Mean satisfaction score measured using the PortionSize Ed User Satisfaction Survey (USS), a 10-item Likert-style instrument that evaluates ease of use and satisfaction with app components including photo features, videos, and feedback. Items are scored on a scale of 1 to 5. The USS also includes open-ended questions for qualitative feedback.
  Units of Measure:
  Score on a 1-5 Likert scale (higher scores indicate greater satisfaction)
  Direction of Scoring:
  Higher scores indicate greater satisfaction and ease of use.
Participant Engagement with the PortionSize Ed App | 11 months
  Mean number of app logins and food photo entries submitted by participants over the 12-week intervention period. Engagement will be assessed using backend app usage data, with higher counts indicating greater engagement.

SECONDARY OUTCOMES:
Mediterranean Diet Adherence Score (MEDAS-14) | 11 months
  Mean change in dietary adherence to the Mediterranean Diet, assessed using the 14-item Mediterranean Diet Adherence Screener (MEDAS-14), a validated questionnaire with scores ranging from 0 to 14. Higher scores indicate better adherence to the Mediterranean Diet.
App-Based Proportion-of-Goal Mediterranean Diet Adherence Score | 11 months
  Mean proportion of Mediterranean Diet food group goals met over the study period, calculated from PortionSize Ed app data. For each tracked food group, participants receive a score from 0 to 1 based on the ratio of actual intake to the goal intake (capped at 1.0). The average across all food groups yields a final adherence score from 0 to 1, with higher values indicating closer adherence to dietary goals.
Change in Hemoglobin A1c (HbA1c) from Baseline to Week 12 | 11 months
  HbA1c will be assessed through a venous blood draw analyzed in a certified clinical laboratory.
Change in Lipid Profile from Baseline to Week 12 | 11 months
  Lipid panel including total cholesterol, HDL-C, LDL-C, and triglycerides will be assessed using venous blood samples analyzed in a certified clinical laboratory.
Change in Systolic and Diastolic Blood Pressure from Baseline to Week 12 | 11 months
  Blood pressure will be measured using a calibrated automated monitor after participants are seated quietly for at least 5 minutes. Two readings will be averaged.
Change in Body Composition Measured by DXA | Baseline and 12 weeks
  Total fat mass (kg), fat mass percentage (%), and fat mass index (kg/m²) measured via dual-energy X-ray absorptiometry (DXA).
Change in Body Fat Percentage Measured by BIA | Baseline and 12 weeks
  Body fat percentage measured by bioelectrical impedance analysis (BIA)
Change in Body Circumference and Volume by 3D Optical Scan | Baseline and 12 weeks
  Measurements include waist circumference and total body volume assessed using a 3D optical scanner.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Undecided